CLINICAL TRIAL: NCT01496937
Title: Exploratory Double-blind Placebo-controlled Study for the Assessment of Pharmacokinetics (PK), Safety, Tolerability, and Pharmacodynamics (PD) of Single Ascending Oral Doses of GLPG0974 in Healthy Subjects
Brief Title: First-in-Human Exploratory Single Ascending Dose of GLPG0974
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0974-CL-101
Record Dates: First submitted 2011-12-16; First posted 2011-12-21 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
MeSH Terms: interventions — 4-(((R)-1-(benzo(b)thiophene-3-carbonyl)-2-methyl-azetidine-2-carbonyl)-(3-chloro-benzyl)-amino)-butyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLPG0974 oral solution (Experimental): GLPG0974 oral solution
  Interventions: Drug: GLPG0974
- Placebo oral solution (Placebo Comparator): Placebo oral solution
  Interventions: Drug: GLPG0974

INTERVENTIONS:
Drug: GLPG0974
  Arms: GLPG0974 oral solution
Drug: GLPG0974
  Arms: Placebo oral solution

SUMMARY:
The purpose of this exploratory first-in-human study is to evaluate the amount of GLPG0974 present in the blood (pharmacokinetics) after single oral doses of GLPG0974 given to healthy subjects.

Furthermore, during the course of the study, safety and tolerability as well as the effects of GLPG0974 on mechanism of action-related parameters in the blood (pharmacodynamics) will be characterized compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The amount of GLPG0974 in plasma over time after a single oral dose
  To characterize the amount of GLPG0974 in plasma over time - pharmacokinetics (PK) - after a single oral dose in healthy subjects

SECONDARY OUTCOMES:
Safety and tolerability
  To evaluate the safety and tolerability of GLPG0974 in comparison with placebo after a single oral dose in healthy subjects in terms of adverse events, physical examinations, vital signs, ECG and lab assessments
Inhibition of CD11b on neutrophils in blood after a single oral dose of GLPG0974
  To characterize the pharmacodynamics (PD) of GLPG0974 by means of inhibition of expression of CD11b on neutrophils after a single oral dose in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV; Wouter Haazen, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Antwerp, Belgium